CLINICAL TRIAL: NCT03485664
Title: Acutely Infected Teeth: To Extract Or Not To Extract?
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gökhan Gürses, Research Assistant, Necmettin Erbakan University
Other Study IDs: NecmettinEU-Dentistry-2
Record Dates: First submitted 2018-03-23; First posted 2018-04-02 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Tooth Extraction Status Nos
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Severe pain on percussion of the relevant tooth was considered as basic criteria when deciding on acute infection phase. The acutely infected teeth were labelled as the study group
  Interventions: Procedure: tooth extraction
- Control Group: The asymptomatic teeth were labelled as the control group
  Interventions: Procedure: tooth extraction

INTERVENTIONS:
Procedure: tooth extraction — tooth extraction

SUMMARY:
This prospective study was performed on 82 participants. Severe pain on percussion of the relevant tooth was considered as basic criteria when deciding on acute infection phase. The acutely infected teeth were labeled as the study group (n=35) and the asymptomatic ones as the control group (n=47). The extractions were done in the usual way. Amount of anesthetic solution used and durations of extractions were recorded.

DETAILED DESCRIPTION:
This research designed as a prospective study between February 2017 and June 2017. An ethical committee approval was obtained (document number 2017/01). The patients were selected among medically healthy volunteers, who referred to us for extraction only one mandibular molar tooth. The informed consents were obtained. Exclusion criteria were smoking, oral contraceptive use, any conditions affecting the immune system, usage of antibiotics in last two weeks and the teeth needed surgical extractions.

A total of 82 patients aged between 15 and 79 years (mean 40.52 ± 15.46) met the study criteria. When deciding on acute infection phase, percussion sensitivity was accepted as the basic criteria. It was defined as severe pain when a dental mirror was dropped about 1 cm above the tooth.

Patients with acutely infected teeth were labeled as "study group" (n = 35) and the asymptomatic patients as "control group" (n = 47). The null hypothesis of the study was "there is no significant difference between the acutely infected and asymptomatic lower molar teeth in terms of the complications that may occur during and after tooth extraction". The level of statistical significance was accepted as 0.05 and SigmaPlot 11.0 (Systat Software, Inc., San Jose, Calif.) program was used for statistical analyses.

Surgical Method All the extractions were performed by the same operator. The investigators used 4% Articaine and 1:100,000 epinephrine HCL as the anesthetic solution. Inferior alveolar nerve (IAN) and buccal nerve (BN) blockages were performed by using 1.5 mL. and 0.5 mL of solution, respectively. If the anesthesia had failed, the same procedure was repeated. The amount of anesthetic solution used for each patient was recorded.

Numbness on the half of the lower lip, and feeling no pain when probing the periodontal space of the target tooth was accepted a successful IAN blockage. Then the BN blockage was performed and the routine extraction was completed. Unless there was a radiographically confirmed granulation tissue, the investigators did not curette the extraction sockets. The investigators also did not package any medications into the wounds or did not suture. A sterile damp gauze was placed tightly on the extraction area and the patients were asked to bite it for 20 minutes. Extraction durations were noted for each patient.

All patients were given postoperative instructions. In the presence of a possible complication, they were asked to apply to our clinic and not to use antibiotics on their own.

Postoperative Evaluation of Systemic Condition The investigators called all the patients on first and second post-extraction days for assessing the systemic signs of fever, fatigue, and shivering.

Postoperative Evaluation of The Extraction Wound If the patients applied with severe pain, The investigators recorded onset time and characteristic of the pain. In the intraoral examination, no granulation tissue as a sign of healing and exposed bare alveolar bone was accepted as alveolar osteitis.

The investigators use SigmaPlot 11.0 (Systat Software, Inc., San Jose, CA) package software programme for statistical analysis. To compare the rates of AO, chi-square test with Yates correction was employed. Shapiro-Wilk normality test was performed on the data for the amount of anesthetic solution used and the duration of extractions. Since the data did not fit the normal distribution, nonparametric Mann Whitney U test was used.

ELIGIBILITY:
Inclusion Criteria:

indication for only one mandibular molar tooth extraction (severe pain on percussion labeled as the study group and asymptomatic ones labeled as the control group)

Exclusion Criteria:

smoking, oral contraceptive use, any conditions affecting the immune system, usage of antibiotics in last two weeks the teeth needed surgical extraction

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were selected among medically healthy volunteers, who referred to the investigators for extraction only one mandibular molar tooth. The informed consents were obtained. Exclusion criteria were smoking, oral contraceptive use, any conditions affecting the immune system, usage of antibiotics in last two weeks and the teeth needed surgical extractions.
  percussion sensitivity is used as separator between two groups.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
diagnosis of alveolaris osteitis | 1-4 days
diagnosis of systemic response | 1-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoğlu, Study Director — Academic Member; Bozkurt Kubilay Işık, Study Chair — Concultant; Gökhan Gürses, Principal Investigator — Care Provider
Locations (1):
- Necmettin Erbakan University, Faculty of dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A total of 82 patients aged between 15 and 79 years (mean 40.52 ± 15.46) met the study criteria. When deciding on acute infection phase, percussion sensitivity was accepted as the basic criteria. It was defined as severe pain when a dental mirror was dropped about 1 cm above the tooth.
  Patients with acutely infected teeth were labelled as "study group" (n = 35) and the asymptomatic patients as "control group" (n = 47). Null hypothesis of the study was "there is no significant difference between the acutely infected and asymptomatic lower molar teeth in terms of the complications that may occur during and after tooth extraction". The level of statistical significance was accepted as 0.05 and SigmaPlot 11.0 program was used for statistical analyses.